CLINICAL TRIAL: NCT06723340
Title: Dermatological Assessment of Primary Dermal Irritability Accumulated, Sensitization, Photoallergy and Photosensitization Under Normal Conditions and When Exposed to Sunlight of a Scar Gel
Brief Title: Dermatological Assessment of Primary Dermal Irritability Accumulated, Sensitization, Photoallergy and Photosensitization of a Scar Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORC-137110_EN24-0262-01_02
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Sensitivity, Contact; Photosensitivity; Phototoxicity
MeSH Terms: conditions — Dermatitis, Contact; Photosensitivity Disorders; Dermatitis, Phototoxic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Scar gel
  Interventions: Device: Scar gel

INTERVENTIONS:
Device: Scar gel — Scar gel (medical device - topical application)

SUMMARY:
Evaluate the potential of Primary Dermal Irritability, Accumulated Dermal Irritability, Dermal Sensitization, Photoallergy and Photosensitization, of health products through the application of Patch Test, proving the safety of the product for topical use. The study will be conducted with a Brazilian sample in which 55 research participants will be included. Depending on the results, the present study may support the claim: dermatologically tested, non-irritating, non-sensitizing, non-photoirritating and non-photosensitizing.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes aged 18 to 70 years;
* Phototypes: I, II, III, and IV (For the phototest trial, only phototypes II and III will be considered);
* Intact skin in the application area;
* Willingness to follow the trial procedures and attend the center on the specified dates and times for medical evaluations and for application and reading of dressings;
* Understanding, consent, and signing of the Informed Consent Form (ICF).

Exclusion Criteria:

* Pregnancy or risk of pregnancy/lactation;
* Use of anti-inflammatory drugs within 30 days and/or immunosuppressive drugs up to three months before selection;
* Immunosuppression due to drugs or active diseases;
* Uncompensated endocrinopathies;
* Personal history of atopy;
* Intense sun exposure or tanning sessions up to 15 days before the evaluation or during the study period;
* Plans to bathe in the sea, pool, or sauna during the study;
* Practice of water sports during the study;
* Dermographism;
* Use of oral or topical treatments with vitamin A acid and/or its derivatives up to one month before the start of the study;
* Aesthetic and/or dermatological treatments on the body within three weeks prior to selection;
* Scheduled vaccination during the study period or within three weeks prior to selection;
* History of sensitization, irritation, or photosensitization to topical products;
* Active skin conditions (local and/or widespread) that could interfere with study results;
* Skin reactivity;
* Use of new medications during the study;
* Previous participation in studies with the same product;
* Congenital or acquired immunodeficiency;
* Clinically significant or current evidence of alcohol or drug abuse;
* Known or suspected history of intolerance to any ingredient in the study product;
* History of non-adherence or unwillingness to adhere to the study protocol;
* Employees of Medcin or the sponsoring company involved in the study, or close family members of an employee involved in the study;
* Other conditions deemed reasonable by the researcher for disqualification from study participation. If applicable, this must be noted in the clinical record.

Exclusion Criteria for the Phototest:

* Previous history of conditions exacerbated or triggered by ultraviolet radiation;
* Use of photosensitizing drugs;
* History or presence of photodermatoses;
* Personal or family history of skin cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Absence | 9 weeks
  Absence of Primary Dermal Irritability Accumulated, Sensitization, Photoallergy and Photosensitization under normal conditions and when exposed to sunlight.

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele Ltda, Osasco, São Paulo, Brazil